CLINICAL TRIAL: NCT05308875
Title: Clinical Study of the Safety and Efficacy of Non-viral Site-directed Integrated PD1-BCMA-CART in Adult Treatment of Relapsed or Refractory Multiple Myeloma
Brief Title: Efficacy and Safety Evaluation of PD1-BCMA-CART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bioray Laboratories (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-BRL-202
Record Dates: First submitted 2022-01-27; First posted 2022-04-04 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: 0.5-2×10^6/kgBW
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD1-BCMA-CART (Experimental): Each subject will accept one of the following dosages of PD1-BCMA-CART cells intravenously (IV) on day 0: 0.5-2*10^6/KgBW.
  Interventions: Biological: PD1-BCMA-CART

INTERVENTIONS:
Biological: PD1-BCMA-CART — Single infusion of PD1-BCMA-CART administered intravenously (i.v.)

SUMMARY:
This trial aims to evaluate the safety and efficacy of PD1-BCMA-CART in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
Using gene editing, chimeric antigen receptors recognizing BCMA were integrated into subject self-derived T cells to obtain a large number of BCMA-CART by in vitro amplification, and BCMA-CART back into the subjects could identify and kill myeloma cells in the subjects.This open-label, dose-escalation study was designed to evaluate the safety and antitumor efficacy of PD1-BCMA-CART in the treatment of relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Have the capacity to give informed consent;
* Confirmed diagnosis of active MM as defined by NCCN and IMWG criteria;
* Have a diagnosis of BCMA+ multiple myeloma (MM), (≥ 5% BCMA+ in CD138+ plasma cells by flow cytometry obtained within 45 days of study enrollment);
* Refractory and relapsed MM patients after > 2 cycles of induction therapy,or,have relapsed or treatment refractory disease following autologous stem cell transplant (ASCT);
* ECOG score=0-2.
* Subjects according with any of the following options:

  * Age≥50;
  * Failure with separation of T cells during autologous CART processing; or,
  * Failure with expansion of autologous CART; or,
  * The proportion of T cells in PBMC <10%; or,
  * Won't benefit from autologous CART therapy because of disease progress.

Exclusion Criteria:

* Pregnant or nursing women; Women of reproductive potential must have a negative serum pregnancy test performed within 48 hours of starting conditioning chemotherapy
* Active infection, HIV infection, syphilis serology reaction positive;
* Active hepatitis B, hepatitis C at the time of screening
* Significant hepatic dysfunction as following, SGOT(serum glutamic-oxaloacetic transaminase)> 5 x upper limit of normal; bilirubin > 3.0 mg/dL;
* Lymphotoxic chemotherapeutic agents within 2 weeks of leukapheresis
* serious mental disorder;
* With severe cardiac, liver, renal insufficiency, diabetes and other diseases;
* Participate in other clinical research in the past three months; previously treatment with any gene therapy products
* Contraindication to cyclophosphamide or fludarabine chemotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 90 days after T cell infusion
  Proportion of patients in whom a response among complete response or partial response, as defined by International Myeloma Working group(IMWG) response criteria , will be observed.

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events as a Measure of Safety and Tolerability | Up to 35 days after T cell infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Duration of persistence of PD1-BCMA-CART | Baseline up to 2 year
  Detect the duration of PD1-BCMA-CART after injection using FACS or Q-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Professor, Principal Investigator — First Affliated Hospital of Zhengzhou University
Locations (1):
- First Affliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No